CLINICAL TRIAL: NCT06593860
Title: Toward a Dysarthria Management Model for Linguistically and Culturally Diverse Groups: Foreign Born Immigrants
Brief Title: Dysarthria Management for Minor Groups
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Yunjung Kim, Principal Investigator, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00003763
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease; Dysarthria
Keywords: speech; mental health; diversity
MeSH Terms: conditions — Parkinson Disease; Dysarthria; Speech; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: A total of 32 dyads of PD participants will be recruited (4 groups of 8 participants in each). The PD participants must be monolingual speakers of Korean living in the United States. Using the waitlist randomized controlled trial (RCT) design, three wait control groups (Groups 2, 3, 4) will serve as untreated comparison groups first, but will serve as intervention groups in the following cycle. The proposed study is divided into two kinds of outcome measures, primary (speech function of PD patients) and secondary (communication participation and well-being of PD patients and their families). Each set of outcome measures will address one of the Specific Aims.
Who Masked: Outcomes Assessor
Masking Description: Due to the interactive nature of rehabilitation, masking the intervention to patients and research investigators is impossible. Therefore, we will blind the separate outcome assessors, who will not be involved in the treatment procedures to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Behavioral, remote speech rehabilitation and counseling (Experimental): Speech therapy will replicate the dose prescribed by many treatment programs including LSVT LOUD, LSVT ARTIC and Be Clear, consisting of 16 sessions of 50-60 minutes duration delivered over four weeks. Participants will also be set 15 to 20 minutes of daily home practice. Family education/training will take place once a week over 4 weeks, including two components: family counseling (30 min) and family conversation training (30 min). Family counseling aims to increase the PD families' knowledge about PD in general and to identify goals and potential solutions to problems which cause emotional turmoil. Family conversation training which aims to increase the PD families' knowledge about PD-related communication problems and to raise awareness of their communication patterns, and to support the development of functional strategies. All activities will remotely occur (using Zoom).
  Interventions: Behavioral: Remote speech rehabilitation
- No Intervention:Waitlist control (No Intervention): No intervention programs (speech therapy, counseling) will be provided.

INTERVENTIONS:
Behavioral: Remote speech rehabilitation — Two types of intervention will be provided via online to 32 dyads of people with Parkinson's disease: (1) speech therapy (PD patients) and (2) family education/training (PD families). Speech therapy will replicate the dose prescribed by many treatment programs including LSVT LOUD, LSVT ARTIC and Be Clear, consisting of 16 sessions of 50-60 minutes duration delivered over four weeks. Participants will also be set 15 to 20 minutes of daily home practice. Family education/training will take place once a week over 4 weeks.
  Arms: Intervention: Behavioral, remote speech rehabilitation and counseling

SUMMARY:
This study develops and conduct a small-scale clinical trial study in which the linguistic and cultural diversity of the participants is considered. Speech therapy and counseling services are provided to both patients with Parkinson's disease and their caregivers.

DETAILED DESCRIPTION:
Attention has been increasingly paid to the "culturally and linguistically diverse (CLD)" communities which typically include dialectal users of English, monolingual and multilingual speakers of minority languages, and bilingual speakers of English and a minority language. However, among these, monolingual speakers of minority languages living in the US have been nearly excluded from dysarthria management. Most of these are first-generation immigrants who are well documented to have limited access to financial and medical services and have poorer health outcomes including communication difficulties. This creates critical health disparities in the field of communication rehabilitation.

This study will (1) examine effects of speech therapy on PD patients' speech acoustics and intelligibility, (2) examine effects of the intervention program on communication participation and well-being of both PD patients and their families. Our primary outcome measures, speech intelligibility and acoustic measures, are hypothesized to show improvements. Acoustic predictors of speech intelligibility are expected to include acoustic vowel space and voice onset time. These hypotheses are based on literature reporting (1) positive changes in speech function after intensive treatment programs focusing on vocal effort and hyperarticulation and (2) language-specific contributors to speech intelligibility in PD. Our secondary outcome measures include (1) communication participation and (2) well-being measures which will be obtained from both PD patients and family members. Based on previous research, the measures are hypothesized to show improved communication participation and well-being in both PD patients and their families following therapy.

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of PD
* No history of other neurological disease
* Native speaker of Korean
* Age between 25 and 85
* Diagnosis of dysarthria secondary to PD from an SLP
* Self-reported typical hearing
* Access to high-speed internet for therapy sessions

Exclusion Criteria:

* A score of 23 or below on the Korean Montreal Cognitive Assessment
* Evidence of voice-speech disorders not-related to PD
* Received speech therapy for PD-related problems in the past one year
* Have no family members to participate in the project.

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Speech Intelligibility Score on a Visual Analogue Scale | Immediately after and 6 months after treatment
  Speech intelligibility will be estimated using the visual analogue scale method. Listeners will rate the degree to which they understood the speech recordings on a continuous line. The two ends will be labeled, totally unintelligible and completely intelligible, respectively. Higher scores indicate more intelligible.
Vowel Space Area (kHz) | Immediately after and 6 months after treatment
  Two acoustic measures will be measured as Primary Outcome. The first one is the size of vowel space area, which has been frequently reported to correlate with speech intelligibility in people with Parkinson's disease.
Speaking Rate (syl/s) | Immediately after and 6 months after treatment
  The second acoustic measures to be included as Primary Outcome is speaking rate. This will be reported as the number of syllables produced in one second.

SECONDARY OUTCOMES:
Dysarthria Impact Profile (DIP) | Immediately after and 6 months after treatment
  DIP is an assessment tool designed to measure the psychosocial impact of dysarthria on affected individuals. It consists of several sections with statements rated on a five-point scale, ranging from "strongly agree" to "strongly disagree." DIP incorporates positively and negatively worded statements with differing scoring schemes. This will be obtained from people with Parkinson's disease. Higher scores indicate greater impact of dysarthria.
Everyday Communication Measure | Immediately after and 6 months after treatment
  Family members will also be asked to rate five different aspects of the PD participant's everyday communication abilities using Everyday Communication Measures on a scale of 1 (poor) to 7 (very good). Example questions include, "how easy is it to understand the speaker?" and "how often does the speaker initiate conversation with you?". This will be obtained from family members of PD participants. Lower scores indicate greater difficulties of everyday communication.
Quality of Family Life Scale | Immediately after and 6 months after treatment
  The Family Quality of Life Scale (FQOL) is a 25-item instrument used to measure several aspects of families' perceived satisfaction in terms of quality of family life (e.g., family interaction, emotional well-being, physical/material well-being, and disability-related support). It uses a 1(very dissatisfied)-5 (very satisfied) Likert scale. Higher scores indicated a better quality of family life.
Perceived Stress Scale | Immediately after and 6 months after treatment
  The Perceived Stress Scale (PSP) will be used for measuring psychological stress. Among the three versions of the PSS, the Korean version of PSS-10 will be used. It uses a 0 (never)-4 (very often) Likert scale. Higher scores indicate more stress.

CONTACTS AND LOCATIONS:
Overall Officials: Yunjung Kim, Principal Investigator — Florida State University
Locations (1):
- Florida State University, Tallahassee, Florida, United States